CLINICAL TRIAL: NCT05565872
Title: Effects of Face-to-face Versus Telematic Supervision During a Community-based Exercise Intervention (Urban Training) Plus Therapeutic Education Programme on Exercise Tolerance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Supervision During a Community-based Exercise Intervention (Urban Training) in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other); Gerencia de Atención Primaria, Madrid (Other Government)
Responsible Party: Principal Investigator, Tamara del Corral Núñez-Flores, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22/126-EC_X_Tesis
Record Dates: First submitted 2022-09-27; First posted 2022-10-04 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Diseases, Obstructive; Respiratory Tract Diseases
Keywords: Exercise Therapy; Telerehabilitation; Exercise Tolerance; Physical Activity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Respiratory Tract Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urban training Intervention + therapeutic education program with face-to-face supervision (Experimental): Patients will be advised to walk in the defined urban trails with face-to-face supervision
  Interventions: Behavioral: Urban training
- Urban training Intervention + therapeutic education program with telematic supervision (Active Comparator): Patients will be advised to walk in the defined urban trails with telematic supervision
  Interventions: Behavioral: Urban training

INTERVENTIONS:
Behavioral: Urban training — A community-based exercise intervention (Urban Training) by using public spaces and urban walkable trails, adapted to each patient needs and capabilities

SUMMARY:
This project plans on a community-based exercise intervention (Urban Training) combined with therapeutic education program, by using public spaces and urban walkable trails, adapted to each patient needs and capabilities in patients with chronic obstructive pulmonary disease (COPD). The main objective of the present study is to evaluate the effects comparing different levels of supervision (face-to-face vs telematic) in the short-, medium- and long-term with respect to: (primary outcome): exercise capacity, and (secondary outcomes): physical activity, quality of life, mental health and COPD exacerbations.

DETAILED DESCRIPTION:
It is a single-blind randomized clinical trial study. Each participant will be randomly assigned to one of the following groups: (1) Urban training Intervention + therapeutic education program with face-to-face supervision, (2) Urban training Intervention + therapeutic education program with telematic supervision

Each exercise training program will be applied once per day, 3 sessions per week during 12 weeks.

The group with Urban training Intervention with face-to-face supervision will be supervised by a physiotherapist once a week. The group with Urban training Intervention with telematic supervision will be supervised by a phone call once a week. To record compliance, participants from all groups were asked to complete a diary at the end of every training session.

The therapeutic education program will consisted of 1 session/week during 4 weeks.

Participants received baseline assessments at the beginning of the intervention, post-intervention assessments at the end of the 13th week, 6 months of follow-up and 12 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* COPD diagnosed by pulmonary function tests during clinical stability, with a ratio of forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ≤ 0.70
* Clinical stability, defined as at least 6 weeks without COPD exacerbation

Exclusion Criteria:

* Neuromuscular or neurological disorders and/or psychiatric or cognitive conditions that hindered they ability to cooperate
* Comorbidity that could interfere with study intervention (e.g., severe orthopaedic problems)
* Previous inclusion in a rehabilitation programme (previous 6 months)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Change in exercise capacity | Baseline, post-intervention (up to 13 weeks), 6 months and 12 months
  Change in exercise capacity between baseline, up to 13 weeks, 6 months and 12 months, as measured by 6-min walking distance

SECONDARY OUTCOMES:
Change in physical activity | Baseline, post-intervention (up to 13 weeks), 6 months and 12 months
  Change in physical activity between baseline, up to 13 weeks, 6 months and 12 months follow-up, as measured during 1 week by accelerometer
Change in quality of life | Baseline, post-intervention (up to 13 weeks), 6 months and 12 months
  Change in quality of life between baseline, up to 13 weeks, 6 months and 12 months follow-up, as measured by COPD Assessment Test
Change in anxiety and depression symptoms | Baseline, post-intervention (up to 13 weeks), 6 months and 12 months
  Change in anxiety and depression symptoms between baseline, up to 13 weeks, 6 months and 12 months follow-up, as measured by the Hospital Anxiety and Depression Scale (HADS), which consists of 14 items divided into 2 subscales for anxiety and depression. Each item is scored on a 4-point Likert scale ranging from 0 to 3, with scores ranging from 0 to 42 and an optimal cut-off score of ≥13.
COPD exacerbations | Post-intervention (up to 13 weeks), 6 months and 12 months
  Number and duration of COPD exacerbations, and admissions to emergency-room or hospital

OTHER OUTCOMES:
The effect of an attendance at an urban training program on changes in self-efficacy | Baseline, post-intervention (up to 13 weeks), 6 months and 12 months
  Changes between baseline, up to 13 weeks, 6 months and 12 months follow-up in self-efficacy measured by the self-efficacy to regulate the exercise scale.
Adherence to treatment | Post-intervention (up to 13 weeks), 6 months and 12 months
  Change in adherence to treatment between post-intervention (up to 13 weeks), 6 months and 12 months follow-up, as measured by the AdT-Physio scale (adherence to physical therapist intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara del Corral, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Zona Básica de Salud Torrejón de Ardoz, Torrejón de Ardoz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Balcells E, Benet M, Borrell E, Celorrio N, Delgado A, Jane C, Marin A, Martin-Cantera C, Monteagudo M, Montella N, Munoz L, Ortega P, Rodriguez DA, Rodriguez-Roisin R, Simonet P, Toran-Monserrat P, Torrent-Pallicer J, Vall-Casas P, Vilaro J, Garcia-Aymerich J. Long-term efficacy and effectiveness of a behavioural and community-based exercise intervention (Urban Training) to increase physical activity in patients with COPD: a randomised controlled trial. Eur Respir J. 2018 Oct 18;52(4):1800063. doi: 10.1183/13993003.00063-2018. Print 2018 Oct. PMID 30166322
- [Background] Arbillaga-Etxarri A, Gimeno-Santos E, Barberan-Garcia A, Benet M, Borrell E, Dadvand P, Foraster M, Marin A, Monteagudo M, Rodriguez-Roisin R, Vall-Casas P, Vilaro J, Garcia-Aymerich J; Urban Training Study Group. Socio-environmental correlates of physical activity in patients with chronic obstructive pulmonary disease (COPD). Thorax. 2017 Sep;72(9):796-802. doi: 10.1136/thoraxjnl-2016-209209. Epub 2017 Mar 1. PMID 28250201